CLINICAL TRIAL: NCT03832790
Title: Sleep, Glycemic Control, and Insulin Resistance in Adolescents With Type 1 Diabetes
Acronym: SunDIAL
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Colorado Clinical & Translational Sciences Institute (Unknown); Ludeman Family Center for Women's Health Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: 19-0186
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Type1diabetes; Adolescent Behavior; Sleep
MeSH Terms: conditions — Adolescent Behavior | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adolescents with type 1 diabetes: Adolescents ages 14-19 with type 1 diabetes
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — observation

SUMMARY:
Despite advancements in care, most adolescents with T1D have higher BMI and significantly higher HbA1c than recommended and are markedly IR, placing them at increased risk for CVD1,2. Thus, alternative approaches to improve and maintain glycemic control, IR, and BMI for adolescents with T1D are urgently needed. This proposal moves beyond the current insulin and carbohydrate counting-focused lifestyle change paradigm to focus on sleep and circadian misalignment, which will allow for identification of new mechanisms that can be directly translated into future intervention and prevention trials. The goal of the current study is to utilize multiple objective measures of sleep duration, timing (actigraphy), and circadian rhythm (melatonin) in adolescents with type 1 diabetes (T1D; N = 40) and examine relationships with glycemic control, IR, vascular health, and BMI. Further, qualitative methodology will be used to identify barriers and facilitators to healthy sleep in adolescents with T1D.

ELIGIBILITY:
Inclusion Criteria:

* attending high school
* diagnosis of type 1 diabetes >1 year

Exclusion Criteria:

* current diagnosis of a sleep disorder (e.g., insomnia, OSA) or abnormal scores on sleep disorders screening measures
* regular use of medications affecting sleep (e.g., stimulants, atypical antipsychotics, melatonin, other sleep aids)
* HbA1c ≥11 or >14% for the previous 2+ measurements
* IQ<70 or severe mental illness

Ages: 14 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescents with type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
HbA1c | at 60 days
  HbA1c
glycemic variability | at 2 weeks
  CGM glucose SD
insulin sensitivity from hyperinsulinemic euglycemic clamp | at study entry (baseline)
  Si
BMI | at study entry (baseline)
  body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus/Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No